CLINICAL TRIAL: NCT05896176
Title: Screening for Obstructive Sleep Apnea Syndrome in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Tania Vanhée, Dr., Université Libre de Bruxelles
Other Study IDs: P2022/377 / CCB B4062022000198
Record Dates: First submitted 2023-04-10; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: child
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Immunologic Memory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric Sleep Questionnaire (PSQ) +: Patient who obtained a score of 7 or more on the PSQ
  Interventions: Diagnostic Test: a clinical examination and anamnesis
- Pediatric Sleep Questionnaire (PSQ) -: Patient who obtained a PSQ score less than 7

INTERVENTIONS:
Diagnostic Test: a clinical examination and anamnesis — The investigators compare the results of the PSQ alone with the elements provided by the clinical examination regarding the referral of patients to the Otolaryngologist (ENT) consultation.
  Groups: Pediatric Sleep Questionnaire (PSQ) +

SUMMARY:
To be able to diagnose obstructive sleep apnea syndrome (OSAS) in a patient, polysomnography (PSG) remains the gold standard. However, this is expensive, involves a considerable workload and is quite complex. Additionally, the wait time from when the patient was referred for PSG to when it is done can take up to 5-6 months. Simpler screening tools have therefore been developed, such as questionnaires. The questionnaires are subjective tools completed by the parents based on the observation of the child's sleep, behavioral problems, etc. These questionnaires have shown usefulness in sorting out patients to be referred to a sleep specialist, an Oto-Rhino-Laryngologist (ENT) or an orthodontist before performing a PSG in view of the difficulty of access to it. The Pediatric Sleep Questionnaire (PSQ) is a tool that was developed by Chervin and his colleagues to screen children with OSAS. This questionnaire is a reliable and scientifically validated tool. In addition, the PSQ is the most accurate questionnaire from a screening point of view. However, the American Academy of Pediatric Dentistry (AAPD) considers that the questionnaires, among others, the PSQ, are not sensitive enough to detect OSAS in a child. They offer an anamnesis as well as a clinical examination to be carried out in addition to the few questions taken from the PSQ that they consider useful for screening patients at risk. The investigators can therefore ask themselves the following question: "Is the PSQ sufficient on its own or do the investigators obtain better results when the investigators carry out a complete anamnesis as well as a clinical examination? "

DETAILED DESCRIPTION:
1. Bibliographic research methodology

   In order to have a relevant bibliographic base, the investigators selected articles with a high level of evidence and the most recent.

   For this, the investigators carried out their research on the following sites and databases: Pubmed, Sciences Direct, Google Scholar, ResearchGate, Tripdatabase and Cible +.

   Several research equations have allowed us to have satisfactory results. When the results were too broad, the investigators restricted their search to meta-analyses and systematic reviews. The following keywords were used: "Pediatric Sleep Questionnaire", "dentistry", "sleep apnea", "child", "surveys and questionnaires", "sleep apnea, obstructive", "diagnosis accuracy"

   The most relevant articles that allowed them to establish the research question were found on Pubmed and Sciences Direct. (appendix n°1) Concerning Google Scholar, Tripdatabase and Cible +, the articles found were either already selected articles or were not sufficiently targeted on the subject.
2. Agreement of the ethics committee

   The study is a prospective observational study carried out within the Erasmus HUB site and therefore required the approval of its ethics committee. The required documents were introduced on the DycoFlow platform on August 31, 2022. They gave their agreement to submit my request to the ethics committee on September 20, 2022. The Erasmus ethics committee gave its agreement on September 9, 2022. December 2022.
3. Study methodology

I. Inclusion and exclusion criteria

The investigators decided to limit the study to children aged 2 to 8 years. Indeed, interceptive orthodontic treatment must be performed before the 9th birthday to be reimbursed if necessary. Moreover, if ENT surgery is necessary (tonsillectomy for example), it is advantageous to perform it as soon as possible. quickly as possible to avoid the long-term consequences of mouth breathing. The investigators also excluded patients whose parents did not speak French.

I. Objective of the study

The study will therefore consist in comparing the results using on the one hand the PSQ only, on the other hand the clinical examination and the anamnesis as well as the three together and see if the results are comparable.

II. Realization of questionnaires

* Pediatric Sleep Questionnaire translated into French (validated translation)
* Anamnesis
* Clinical examination

Concerning the anamnesis and the clinical examination, the investigators based themselves on the recommendations given by the AAPD. Indeed, some studies have shown that the questionnaire gives better results when combined with a clinical examination.

III. Data collection

The study took place within the Erasmus site HUB, at the Erasmus Medical Center (EMC) during pediatric dentistry consultations.

The parents of the patients were approached from the beginning of the consultation in order to integrate the study. Oral explanations concerning the purpose and conduct of the study were given in addition to informed consent. In addition, the children also received appropriate informed consent explaining the course of the study if the age and maturity of the child permitted it.

The PSQ and the anamnesis are carried out during the consultation with the parent. Once the consultation is over, the clinical examination is carried out with the consent of the child.

If the PSQ turned out to be positive, i.e. the child obtained a score equal to or greater than 7 positive responses out of 22, a liaison letter was sent to refer the child to an ENT specialist. The investigators also asked for an e-mail report of the consultation. This was also the case for the anamnesis and the clinical examination.

ELIGIBILITY:
Inclusion Criteria:

- 2-8 years

Exclusion Criteria:

* Patients who do not speak French

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients between 2 and 8 years old presenting to the pediatric dentistry consultation at Erasmus Hospital,EMC site, speaking French and agreeing to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
PSQ + or - | The data collection is carried out during the consultation
  Patient positive or negative on Pediatric Sleep Questionnaire (PSQ)
History/clinical examination + or - | The data collection is carried out during the consultation
  Patient positive or negative at History/clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Fairouz Ben Abdelouahed, Principal Investigator — Directrice du service de Dentisterie HUB
Locations (1):
- Tania Vanhée, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No